CLINICAL TRIAL: NCT07075926
Title: Evaluation of Left Ventricular Function to Predict Weaning Success in the Intensive Care Unit: A Prospective Observational Study
Brief Title: Evaluation of Left Ventricular Function to Predict Weaning Success in the Intensive Care Unit
Status: Recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: Weaning-Left Heart
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Weaning Failure of Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Weaning Candidates: This group includes adult ICU patients who are receiving mechanical ventilation and have met standardized weaning criteria. All patients in this cohort will undergo transthoracic echocardiographic (TTE) assessment before extubation, without any experimental intervention applied.
  Interventions: Diagnostic Test: Echocardiographic Assessment

INTERVENTIONS:
Diagnostic Test: Echocardiographic Assessment — All participants will receive a standardized transthoracic echocardiographic (TTE) examination within 2 hours after meeting weaning criteria. The following cardiac function parameters will be recorded:
  LVOT Velocity Time Integral (VTI)
  Mitral Annular Plane Systolic Excursion (MAPSE)
  E/e' ratio
  E/A ratio
  Mitral Deceleration Time (MDT)
  Myocardial Performance Index (Tei index)
  The echocardiographic data will be used to investigate the association between left ventricular function and weaning success.

SUMMARY:
The goal of this prospective observational study is to evaluate whether left ventricular function parameters assessed via transthoracic echocardiography (TTE) can predict weaning success from mechanical ventilation in adult intensive care unit (ICU) patients. The main questions it aims to answer are:

Can the Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI) predict successful extubation?

What is the prognostic value of other echocardiographic measures such as Mitral Annular Plane Systolic Excursion (MAPSE), E/e' ratio, E/A ratio, Mitral Deceleration Time (MDT), and Myocardial Performance Index (Tei index) in forecasting weaning outcomes?

Participants will:

Be adults receiving mechanical ventilation and scheduled for weaning

Undergo transthoracic echocardiography (TTE) within 2 hours after meeting weaning criteria

Have the following parameters measured: LVOT VTI, MAPSE, E/e', E/A, MDT, and Tei index

Be monitored for 24 hours post-extubation to determine if they remain off ventilatory support, including reintubation, non-invasive ventilation, or high-flow oxygen therapy

This study aims to provide a comprehensive understanding of how systolic, diastolic, and global cardiac functions influence extubation success, potentially improving ICU decision-making and reducing complications, length of stay, and healthcare costs.

DETAILED DESCRIPTION:
This prospective, single-center observational study aims to assess the predictive value of left ventricular function parameters obtained via transthoracic echocardiography (TTE) in determining weaning success in mechanically ventilated adult ICU patients.

Following fulfillment of weaning criteria, patients will undergo TTE evaluation within 2 hours. The echocardiographic assessment will include the measurement of:

Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI)

Mitral Annular Plane Systolic Excursion (MAPSE)

E/e' ratio

E/A ratio

Mitral Deceleration Time (MDT)

Myocardial Performance Index (Tei index)

These measurements aim to reflect systolic, diastolic, and global left ventricular functions. After the echocardiographic assessment, patients will be followed for 24 hours to determine weaning success, defined as the ability to maintain spontaneous breathing without reintubation, non-invasive ventilation, or high-flow oxygen support.

By integrating non-invasive, bedside cardiac function assessments into the extubation decision-making process, the study seeks to contribute to more physiologically guided weaning strategies. The results may help reduce weaning-related complications and optimize resource use in critical care settings

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving mechanical ventilation in the ICU
* Planned extubation after meeting standard weaning criteria
* Hemodynamically stable at the time of echocardiographic evaluation
* Written informed consent obtained from the patient or legally authorized representative

Exclusion Criteria:

* Surgery within the previous 24 hours
* Presence of significant valvular heart disease or known cardiomyopathy
* Inadequate acoustic window for transthoracic echocardiography
* Ongoing use of extracorporeal support (e.g., ECMO)
* Patients with Do-Not-Resuscitate (DNR) orders or expected to die within 24 hours
* Re-intubation planned prophylactically regardless of clinical status
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients admitted to the intensive care unit (ICU) who are receiving invasive mechanical ventilation and are scheduled for extubation after fulfilling standard weaning criteria. All participants will be hemodynamically stable at the time of echocardiographic assessment. Patients with significant structural heart disease, inadequate echocardiographic imaging windows, or ongoing extracorporeal support will be excluded. The population represents a typical critically ill cohort undergoing weaning from mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07-15 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of LVOT VTI in Determining Weaning Success | Within 24 hours after extubation
  To evaluate whether the Left Ventricular Outflow Tract Velocity Time Integral (LVOT VTI) measured by transthoracic echocardiography (TTE) within 2 hours after fulfilling weaning criteria can predict successful weaning from mechanical ventilation. Successful weaning is defined as maintaining spontaneous breathing for at least 24 hours without requiring reintubation, non-invasive ventilation, or high-flow nasal oxygen therapy.

SECONDARY OUTCOMES:
Predictive Value of Additional Left Ventricular Function Parameters in Weaning Success | Within 24 hours after extubation
  To assess whether echocardiographic parameters other than LVOT VTI - including Mitral Annular Plane Systolic Excursion (MAPSE), E/e' ratio, E/A ratio, Mitral Deceleration Time (MDT), and Myocardial Performance Index (Tei index) - are associated with successful weaning from mechanical ventilation. These parameters reflect systolic, diastolic, and global left ventricular function and will be measured using transthoracic echocardiography prior to extubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)